CLINICAL TRIAL: NCT07252479
Title: A Multi-center, Open-label, Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of AN9025 in Participants With Advanced or Metastatic Solid Tumors Harboring RAS Mutations
Brief Title: Evaluation of RAS Inhibitor Treatment in Participants With Advanced or Metastatic Solid Tumors Harboring RAS Mutations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adlai Nortye Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN9025S0101
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors (Phase 1); RAS Mutation
Keywords: RAS; RAS (ON); RAS Solid Tumor; KRAS G12X(C/D/V); KRAS G13D; NRAS Q61X(L/K); Oral Pan RAS medication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AN9025 Treatment (Experimental): Oral administration of AN9025 capsules
  Interventions: Drug: AN9025 oral capsule

INTERVENTIONS:
Drug: AN9025 oral capsule — AN9025 is a novel, oral, small molecule pan-RAS (ON) inhibitor that binds cyclophilin A (CypA) with a slow dissociation rate, forming a tri-complex with guanosine triphosphate (GTP) bound state of both mutant and wild-type RAS proteins. AN9025 exhibits potent anti-proliferative activity in RAS-addicted cancer cell lines, demonstrates favorable pharmacokinetics (PK), pharmacodynamics and an acceptable tolerability profile in vivo.

SUMMARY:
The goal of this clinical trial is to learn determine if AN9025 is safe and tolerable to treat solid cancer tumors with specific genetic mutations. It will help identify doses for use in future testing and establish the safety profile of the drug. The main questions it aims to answer are:

Which dose(s) of AN9025 are safe and tolerable for use in evaluating anti-tumor activity in participants with Rat Sarcoma oncogene (RAS) mutated solid tumors? What medical problems do participants have when taking AN9025?

Participants will:

Take AN9025 by mouth every day until their disease progresses, they experience severe ill side effects from taking the drug, or withdraw from the study due to their own choice or as recommended by their physician.

Visit the clinic 3-4 times during the first 21 days of treatment for study testing, blood draws and tumor tissue sample collection (if needed). The blood draws will be used to check drug levels in the participants blood for research purposes.

Visit the clinic every 21 days for checkups and tests and monitoring of participant progress.

Return to the clinic at 14 and 30 days after AN9025 treatment is stopped. Participants will be contacted every 3 months to check on the participants disease status and general well being.

Participants may also partake in a food effect study, where the effect of eating is studied to see if there is any effect on AN9025 in the body.

DETAILED DESCRIPTION:
This is a first-in-human, open label, multi-center, multiple-ascending dose escalation, phase I study consisting of three parts: Part 1 Dose-Escalation, Part 2 Food Effect Assessment and Part 3 Dose-Expansion (See Figure 1, Figure 2, Figure 3 and Figure 4). The study is designed to evaluate the safety, tolerability, PK, and preliminary efficacy of AN9025, an oral pan-RAS (ON) inhibitor, in participants with advanced or metastatic solid tumors that harbor RAS mutations. In addition, the effect of food intake on the PK of AN9025 will be preliminarily investigated. The study will be conducted in the United States and China.

Part 1 Dose-Escalation is designed to identify the Maximum Tolerated Dose (MTD) and/or Recommended Dose for Expansion (RDE) in participants with advanced or metastatic RAS-mutant solid tumors. Participants will be evaluated for Dose-limiting Toxicities (DLTs) in escalating dose and back fill cohorts. Participants enrolled in escalating dose cohorts will receive AN9025 with continuous once daily (QD) dosing in 21-day cycles. Participants enrolled in back fill cohorts will start with a single lead-in dose of AN9025 at least 5 days prior to initiating continuous QD dosing to enable PK sampling during the Single-Dose Lead-in period (Cycle 0). Following the Lead-in period, back fill participants will begin Cycle 1 Day 1 of the standard QD 21-day cycle treatment (Figure 3 A).

Part 2 Food Effect Assessment will employ a single-sequence, two-period crossover design in at least 6 participants. Participants will begin with a Food Effect Lead-in period (Cycle 0), receiving a single-dose of AN9025 (at a selected dose level lower than the MTD) under fasting condition, followed by PK sample collection and a washout period. A second single-dose will then be administered under fed conditions, with additional PK sampling and another washout period. Upon completing this lead-in period, participants will transition to the main study treatment, initiating QD dosing from Cycle 1 Day 1 in 21-day cycles (Figure 3 B).

Part 3 Dose-Expansion will evaluate the clinical activity of AN9025 in up to two RAS-mutated solid tumor indications using up to two dose levels selected based on the MTD/RDE established during dose escalation. This phase will further characterize the safety, tolerability, and PK of AN9025 in selected tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old at the time of informed consent.
2. Able to provide informed consent voluntarily before any study-related activities and according to local guidelines.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Have an estimated life expectancy ≥ 12 weeks, in the judgment of the Investigator.
5. Have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic with progression after treatment with available standard therapies.
6. Documentation of KRAS/NRAS/HRAS mutation determined by validated local testing of tumor tissue or circulating free DNA (cfDNA) in a certified laboratory.
7. Have consented to provide archival tumor tissue collected within 5 years or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
8. Part 1 Dose-Escalation and Part 2 Food Effect Assessment: cancers including, but not limited to:

   1. Pancreatic ductal adenocarcinoma (PDAC)
   2. Colorectal cancer (CRC)
   3. Non-small cell lung cancer (NSCLC)
   4. Cutaneous melanoma
   5. Biliary tract cancer (BTC)
9. Part 3 Dose-Expansion:

   Cohort 3A: RAS-mutated solid tumors (2L/3L)
   1. Histologically or cytologically confirmed advanced or metastatic disease
   2. Participants must not have tumors previously tested positive for targetable oncogenic driver mutations including Epidermal Growth Factor Receptor (EGFR), Anaplastic Lymphoma Kinase (ALK), B-Rapidly Accelerated Fibrosarcoma (BRAF), RET, and ROS1
   3. Participants must have received 1 or 2 prior lines of systemic therapy which include prior immune checkpoint inhibitor and platinum chemotherapy administered either concurrently or sequentially, and have not received docetaxel previously
   4. Participants must be refractory to anti-PD-1/PD-L1 therapy.
   5. Adjuvant therapy or multimodal therapy with curative intent is considered prior therapy if disease progression occurred or treatment completion was within 6 months of first dose of AN9025.
   6. Participants must not have tumors previously tested positive for Class I BRAF mutations i.e. V600X.
10. Have adequate organ functions prior to enrollment:

    1. ANC: >= 1.5 x 10^9/L
    2. Platelets: >= 100x 10^9/L
    3. Hemoglobin: >= 9.0 g/dL
    4. AST and ALT: <= 2.5 x Upper Limit of Normal (ULN) or ,+ x ULN if liver metastases are present
    5. Total bilirubin: <= 1.5 x ULN
    6. Creatinine clearance (CrCl): CrCl >= 50 ml/min as determined by Cockcroft-Gaulat formula
    7. International Normalized Ratio (INR) or prothrombin (PT) time or activated partial thromboplastin time (aPTT): PT or aPTT <= 1.5 x ULN or INR < 1.5
11. Have discontinued all previous treatments for cancer with resolution of any adverse events (AEs) to ≤ Grade 1 (except for alopecia, and endocrinopathies that are managed with replacement therapy), and all clinically significant toxicities from prior locoregional therapy, surgery, radiotherapy, or systemic anticancer therapy to ≤ Grade 1 prior to enrollment.
12. Corrected QT interval (QTc) ≤ 470 msec for females and ≤ 450 msec for males per the Fridericia's Formula (QTcF).
13. Able to swallow oral medication and comply with study requirements.
14. Left ventricular ejection fraction (LVEF) greater than 50% on echocardiography or multiple gated acquisition (MUGA) scan.
15. Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for 180 days after the last study treatment administration. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative pregnancy test ≤ 14 days prior to the first dose of the study treatment.

Exclusion Criteria:

Participants meeting any of the following criteria will not be eligible for participation in the study.

1. Are currently enrolled in a clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Have tumors previously tested positive for Class I BRAF mutations i.e. V600X.
3. Prior treatment with a pan-RAS(ON) inhibitor.
4. Gastrointestinal conditions that may interfere with drug absorption (e.g., malabsorption syndrome, chronic nausea/vomiting, active inflammatory bowel disease).
5. Have a serious concomitant systemic disorder that, in the judgment of the Investigator, would compromise the participant's ability to adhere to the protocol, such as the following:

   1. Known human immunodeficiency virus (HIV) infection per HIV 1 and/or 2 antibodies.
   2. Participants with evidence of active Hepatitis B or Hepatitis C infections (positive for Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody)
   3. Active tuberculosis, fungal infection
   4. Active infection requiring intravenous antibiotic therapy. Use of oral antibiotics for minor infections (e.g., uncomplicated UTI or URI) is permitted if clinically stable, at the Investigator's discretion
6. The participant has a serious pre-existing medical condition(s) that, in the judgment of the Investigator, would preclude participation in this study, including interstitial lung disease (ILD), severe dyspnea at rest, or requiring oxygen therapy.
7. Prior or second concurrent primary malignancies that, in the judgment of the Investigator, may affect the interpretation of results. Participants with carcinoma in situ of any origin and participants with prior malignancies who are in remission and whose likelihood of recurrence is very low (such as basal cell carcinoma), as judged by the Investigator, or malignancies that don't need treatment (i.e., small renal cell carcinoma [RCC] and localized prostate cancer) are eligible for this study.
8. Moderate or severe cardiovascular disease, such as the following:

   1. congestive heart failure
   2. New York Heart Association Class III/IV heart disease
   3. unstable angina pectoris
   4. myocardial infarction or cardiovascular event within the last 6 months before enrollment
   5. valvulopathy that is severe, moderate, or deemed clinically significant
   6. arrhythmias that are symptomatic or require treatment (not including Participants with rate-controlled supraventricular tachycardia)
   7. a history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT syndrome)
   8. require the use of concomitant medications that prolong the QT/QTc interval
9. Have symptomatic central nervous system (CNS) malignancy or metastasis.
10. Are pregnant or planning to become pregnant during the study or within 6 months following the last dose of AN9025. Plan to be breastfeeding from the initial dose of study treatment or within 6 months following the last dose of AN9025.
11. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
12. Use of other herbal supplements, traditional medicines, or prescription medications that are known or suspected to interact with the investigational product or effect disease treatment/side effect management, as determined by the study Investigator.
13. Known allergic reaction against any of the components of the study treatments.
14. Current use of drugs known to be strong or moderate inhibitors or inducers of isoenzyme cytochrome P450 3A4 (CYP3A4) including herbal medications.
15. Current use of drugs known to be of P-glycoprotein (P-gp) inhibitors.
16. Participants who are unable to discontinue proton pump inhibitors (PPIs) for at least 5 days prior to the first dose of AN9025, or unable to abstain from PPI use throughout the study treatment period.
17. Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and Investigator's knowledge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
• Nature and frequency of dose limiting toxicities (DLTs) | 21 days after first dose
  • Incidence, nature, and severity of adverse events according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Preliminary anti-tumor activity:Objective response rate (ORR) | Tumor assessments will occur at baseline and then every 6 weeks starting from Cycle 3, Day 1 up to Cycle 9, Day 1 and then every 12 weeks thereafter (± 1 week window), through study completion, for an average duration of 1 year
  • Measure the Objective response rate (ORR)
• Characterization of the PK profile of AN9025 following administration as an oral capsule formulation | At time points pre-dose, 1, 2, 4, 6, 8, 24 hours post dose
  • The assessment will include, but not limit to, the following PK parameters for AN9025
  - AUC(inf) after single dose and AUC (0-τ) after single and multiple doses Maximum blood concentration (Cmax)
•Characterization of the PK profile of AN9025 following administration as an oral capsule formulation: steady state characterization | At time points pre-dose, 1, 2, 4, 6, 8, 24 hours post dose
  Accumulation ratio (AR) at steady-state
Characterization of the PK profile of AN9025 following administration as an oral capsule formulation: drug level characterization in blood | At time points pre-dose, 1, 2, 4, 6, 8, 24 hours post dose
  Apparent clearance (CL/F) after single and multiple doses
Characterization of the PK profile of AN9025 following administration as an oral capsule formulation | At time points pre-dose, 1, 2, 4, 6, 8, 24 hours post dose
  AN9025 apparent terminal half-life (t1/2)
Characterization of PK profile of AN9025 following administration as an oral capsule formulation: blood concentration characteristics | At time points pre-dose, 1, 2, 4, 6, 8, 24 hours post dose
  Time to maximum blood concentration (Tmax)
Preliminary anti-tumor activity: disease control rate (DCR) | Tumor assessments will occur at baseline and then every 6 weeks starting from Cycle 3, Day 1 up to Cycle 9, Day 1 and then every 12 weeks thereafter (± 1 week window), through study completion, for an average duration of 1 year
  measurement of the disease control rate (DCR)
Preliminary anti-tumor activity for tumor response | Tumor assessments will occur at baseline and then every 6 weeks starting from Cycle 3, Day 1 up to Cycle 9, Day 1 and then every 12 weeks thereafter (± 1 week window), through study completion, for an average duration of 1 year
  meausrement of the duration of response (DoR)
Preliminary anti-tumor activity: participant survival | Tumor assessments will occur at baseline and then every 6 weeks starting from Cycle 3, Day 1 up to Cycle 9, Day 1 and then every 12 weeks thereafter (± 1 week window), through study completion, for an average duration of 1 year
  Measurement of the participant's progression-free survival (PFS) as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Investigator

OTHER OUTCOMES:
The identification of potential predictive biomarkers associated with response or resistance to AN9025 | Measured at baseline and evaluated at study completion, estimated at 2 years of first enrolled participant.
  • Correlation of clinical outcomes with biomarkers to specific RAS mutation subtypes, and co-mutations in tumor tissue at baseline and progressive disease.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - University of Texas MD Anderson Cancer Center, Houston, Texas